CLINICAL TRIAL: NCT01153204
Title: Satisfaction With the Treatment, Confidence and Naturalness in Engaging in Sexual Activity in Men With Psychogenic Erectile Dysfunction: Randomized Controlled Trial of Three Therapeutic Approaches.
Brief Title: Satisfaction, Confidence and Naturalness in Men With Psychogenic Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DE Satisfaction - 2010
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Group Psychotherapy; Sildenafil [Substance Name]; Patient Satisfaction; Efficacy; Randomized Controlled Trial [Publication Type]
MeSH Terms: conditions — Erectile Dysfunction; Patient Satisfaction | interventions — Psychotherapy, Group; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Psychotherapy (GP) (Experimental): Time-limited group psychotherapy is a technique based on psychodrama, an in-depth method of group psychotherapy. Active methods are used to enable past, present, and future life events to be explored. Sexual issues and their possible solutions are enacted rather than simply discussed. Time-limited group psychotherapy focuses on a central or core issue or a circumscribed area of conflict (psychogenic erectile dysfunction) as the only or major object of intervention efforts.
  Interventions: Behavioral: Group Psychotherapy
- Sildenafil (Active Comparator): Participants took sildenafil citrate 50 mg as needed for sexual activity (on demand), no more than once daily, according to psychiatric prescription. Sildenafil citrate was taken with a glass of water on an empty stomach (at least 2 hours after eating). Participants met with a psychiatrist every month for 30-minutes to report adverse effects and to obtain the following month's dosage of four pills.
  Interventions: Drug: Sildenafil citrate
- Group Psychotherapy (GP) plus Sildenafil (Active Comparator): The same as above.
  Interventions: Other: Group Psychotherapy plus Sildenafil citrate

INTERVENTIONS:
Behavioral: Group Psychotherapy
  Arms: Group Psychotherapy (GP)
Other: Group Psychotherapy plus Sildenafil citrate
  Arms: Group Psychotherapy (GP) plus Sildenafil
Drug: Sildenafil citrate
  Arms: Sildenafil

SUMMARY:
Context and Objectives: Erectile dysfunction severely compromises not only sexual satisfaction, which is well known to be closely linked to overall life satisfaction but is also associated with a lower quality of life, lower self-esteem, depression, anxiety and adverse effects on interpersonal relationships. The objective was to assess the efficacy of psychotherapy and/or sildenafil for psychogenic erectile dysfunction.

Design and Settings: randomized controlled single-blind trial performed at Institute of Psychiatry of the Medical School of at Universidade de São Paulo, São Paulo, Brazil Methods: Thirty patients with mild and moderate psychogenic erectile dysfunction (ED) were randomized to receive for six months: group psychotherapy (GP) plus 50mg sildenafil on demand, or 50mg sildenafil exclusively, on demand, or GP exclusively. Changes in score from baseline for three questions of the Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) were evaluated at end-point and after 3-months follow-up.

Results: satisfaction with the treatment, confidence and naturalness increased in GP plus sildenafil and GP exclusively groups (p=0.001) from baseline to endpoint. The treatment-by-time comparison was not significant at end point versus 3-month follow-ups, in the three groups. No difference was observed in the sildenafil group in the three study periods (P >0.05) Conclusions: Patients with mild and moderate psychogenic ED had higher treatment satisfaction, confidence and naturalness in engaging in sexual activity when receiving GP plus sildenafil or GP exclusively, when compared with sildenafil exclusively, as assessed by these three EDITS questions after 6-months treatment

ELIGIBILITY:
Inclusion Criteria:

1. exclusive diagnosis of psychogenic ED, using a checklist for DSM-IV criteria.Morning erections, situational erections (masturbatory or with another partner), or acute onset are characteristics of psychogenic ED;
2. age between 25 and 50 years;
3. mild and moderate erectile dysfunction according to the International Index of Erectile Function (IIEF);
4. stable heterosexual relationship for at least 1 year, and in accordance with inclusion criteria during short-time psychotherapy focused on sexuality; (f) informed consent from the patient.

Exclusion Criteria:

Patients were excluded if presenting significant clinical diseases, major depressive disorder or other severe mental disorder, primary no erectile sexual disorder (e.g., hypoactive sexual disorder), penile anatomic defects; users of medications that could interfere with sexual function; patients with any kind of physical limitations for the use of sildenafil citrate (current use of nitrates, past history of retinitis pigmentosa, allergies); and significant drug, alcohol or tobacco use

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the treatment
  Changes in scores of EDITS question 1 (satisfaction with the treatment), from baseline to endpoint and 3-months follow-up in the three groups.

SECONDARY OUTCOMES:
Confidence in engaging in sexual activity
  Changes in EDITS questions 7 (confidence in engaging in sexual activity) evaluated in three study periods: baseline, end-point and 3-months follow-up in the three groups.
Naturalness in engaging in sexual activity
  Changes in EDITS questions 11 (naturalness in engaging in sexual activity), evaluated in three study periods: baseline, end-point and 3-months follow-up in the three groups.

REFERENCES:
- [Derived] Melnik T, Abdo CH, de Moraes JF, Riera R. Satisfaction with the treatment, confidence and 'naturalness' in engaging in sexual activity in men with psychogenic erectile dysfunction: preliminary results of a randomized controlled trial of three therapeutic approaches. BJU Int. 2012 Apr;109(8):1213-9. doi: 10.1111/j.1464-410X.2011.10516.x. Epub 2011 Aug 22. PMID 22455403